CLINICAL TRIAL: NCT01652131
Title: Colloid Volume Kinetics in Morbidly Obese Patients Under General Anaesthesia
Brief Title: Behaviour of Intravenous Solutions in Obese Patients Under General Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Medical Sciences and Nutrition, Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Maria Victoria Hernandez Martinez, M.D., National Institute of Medical Sciences and Nutrition, Salvador Zubiran
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: REF.343
Record Dates: First submitted 2012-07-25; First posted 2012-07-27 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Obesity; Obesity, Morbid
Keywords: general anesthesia; volume kinetics
MeSH Terms: conditions — Obesity; Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tetrastarch (130/0.4) (Other): In obese patients candidates to laparoscopic gastrojejunal bypass an infusion of Tetrastarch (130/0.4)) of 15mL/kg (of corrected weight) will be initiated after protocoled induction of general anesthesia. Blood samples will be taken at time 0 (after induction of anesthesia and before initiating infusion) and then every 5 minutes for half an hour and then every 15 minutes up to 90 minutes. Blood samples will be processed in the Institution's laboratory. Urine will be measured at the end of the intervention. With these data kinetic parameters will be estimated for each patient.
  Interventions: Other: Tetrastarch (130/0.4)

INTERVENTIONS:
Other: Tetrastarch (130/0.4)
  Other Names: Voluven 6%

SUMMARY:
There is no objective evidence of how long intravenous solutions remain inside venous blood vessels after they have been administered, therefore there is no definite guideline of how to administer them in the preoperative setting. Besides, obese patients represent a particular group of subjects as they theoretically with-hold a constant inflammatory response and that would modify the way solutions behave intravenously, that is how long they remain inside.

Having said this, we wish to describe the way colloid solutions behave in this group of patients by taking serial blood samples in 12 obese patients after a colloid infusion, to calculate plasma dilution curves based on hemoglobin dilution and therefore infer the time it remains intravascularly.

All this in the hope this information will help, in the near future, to establish a more objective way to use these solutions and avoid possible complications due to over-administration.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of obesity (IMC >35kg/m2) that will be treated with gastrojejunal laparoscopic bypass

Exclusion Criteria:

* Renal failure KDOQI >3
* Cardiac failure NYHA III-IV
* Sepsis
* Allergy to tetrastarch
* Allergy to any of the anesthetic medication that is to be used in the protocol previously established
* Patients in which vasoactive drugs are used
* Patients in which the blood samples are completed.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2012-05; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
description of colloid volume kinetics in obese patients after the infusion of Tetrastarch (130/0.4) | 90 minutes after beginning of the infusion
  different kinetic parameters will be used to asses the behavior of the colloid solution

CONTACTS AND LOCATIONS:
Overall Officials: Miguel F Herrera Hernandez, MD MSc PhD, Study Director — National Institute of Medical Sciences, Salvador Zubiran; Maria V Hernandez Martinez, M.D., Principal Investigator — National Institute of Medical Sciences, Salvador Zubiran
Locations (1):
- National Institute of Medical Sciences, Salvador Zubiran, Mexico City, Mexico City, Mexico